CLINICAL TRIAL: NCT06757543
Title: A Stepped Wedge Cluster Randomised Trial of Video Versus Direct Laryngoscopy for Intubation of Newborn Infants
Acronym: NEU-VODE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College Dublin (Other)
Collaborators: National Maternity Hospital, Ireland (Other); Leiden University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEU-VODE 01
Record Dates: First submitted 2024-12-20; First posted 2025-01-03 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Intubation; Intubation Complications; Infant, Newborn; Infant Respiratory Distress Syndrome; Video Laryngoscopy
Keywords: infant, newborn; video laryngoscopy; intubation; stepped wedge cluster randomised trial
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Intervention Model Description: Stepped wedge cluster randomised study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Video laryngoscopy (Experimental): Participant intubated during period where first intubation attempt routinely made with video laryngoscope
  Interventions: Device: Video laryngoscopy
- Direct laryngoscopy (Active Comparator): Participant intubated during period where first intubation attempt routinely made with standard laryngoscope
  Interventions: Device: Direct laryngoscopy with standard laryngoscope

INTERVENTIONS:
Device: Video laryngoscopy — Video laryngoscopy with C-MAC (Karl Storz, Tuttlingen, Germany)
  Arms: Video laryngoscopy
Device: Direct laryngoscopy with standard laryngoscope — Direct laryngoscopy with standard laryngoscope
  Arms: Direct laryngoscopy

SUMMARY:
Many newborn babies have difficulty breathing. When babies need a lot of help, a doctor will intubate them - i.e. put a tube into their windpipe (trachea) - so that they can be given support with a breathing machine. Intubation is a difficult procedure, during which many babies have falls in their blood oxygen levels and heart rate. When doctors intubate babies, they use a device called a laryngoscope to identify the entrance to the windpipe. A standard laryngoscope has a light at its tip. When doctors use this device, they insert it into the baby's mouth and then look directly into the mouth to find the entrance (direct laryngoscopy). Less than half of first attempts to insert a tube are successful using this device. More recently, video laryngoscopes have been developed. These devices also have a camera at the tip and display a magnified view of the entrance to the windpipe on a screen. A study at one hospital showed that the doctors there inserted the tube at the first attempt more often when they used a video laryngoscope instead of a standard laryngoscope. This study was not large enough to see whether fewer babies had low oxygen levels or heart rate during the procedure.

The goal of this clinical trial is to see whether more newborn babies are intubated at the first attempt without falls in their blood oxygen levels or heart rate when the doctors use video laryngoscopy compared to direct laryngoscopy.

Hospitals where doctors routinely intubate babies by looking directly into the mouth will take part in the NEU-VODE study. From the start of the study, the doctors at each hospital will continue with their usual approach to intubation and collect information about intubation attempts. As the study progresses, the doctors at each participating hospital will switch one--by-one to routinely attempting intubation with a video laryngoscope. The date on which they switch will be determined by chance. By the end of the study, each hospital will have had a study period where babies were routinely intubated using direct laryngoscopy and video laryngoscopy.

At the end of the study, the information collected from all the babies intubated during the study will be compared to see if more babies were successfully intubated at the first attempt without falls in their blood oxygen levels or heart rate in the video laryngoscopy group.

DETAILED DESCRIPTION:
INTRODUCTION Many newborn infants have difficulty breathing after birth. Some of these babies have a tube inserted into their "windpipe" (trachea) - an endotracheal tube (ETT) - through which they are given breathing support (ventilation). When clinicians attempt to intubate (insert an ETT), they use an instrument called a laryngoscope to view the airway in order to identify the entrance to the trachea (larynx). Standard laryngoscopes have a "blade" (which, despite its name, is not sharp) with a light at the tip. Doctors insert the blade into the baby's mouth to view the larynx. Traditionally, clinicians used a standard laryngoscope to look directly into the baby's mouth to view the larynx (direct laryngoscopy, DL). When clinicians attempt to intubate newborns with DL, less than half of first attempts are successful. Also adverse effects - such as falls in the blood oxygen levels (fall in oxygen saturation (SpO2), or "desaturation"), slowing down of the heart rate (bradycardia), oral trauma - are relatively common.

In recent years, video laryngoscopes (VL) have been developed. In addition to a light, VL have a video camera at the tip of the blade. This camera acquires a view of the larynx and displays it on a screen that the clinician views when attempting intubation (indirect laryngoscopy). In a randomised study performed at the National Maternity Hospital, Dublin, Ireland, more infants were successfully intubated at the first attempt when clinicians used VL compared to DL [79/107 (74%) versus 48/107 (45%), P<0.001]. While this study was large enough to show that VL resulted infants being successfully intubated at the first attempt in one hospital, it couldn't give information about how it might work in a range of hospitals, and it wasn't large enough to see what effect VL had on adverse events. There is a large difference in cost between a standard laryngoscope (approx. €300) and a video laryngoscope (approx. €21,000). This is a matter of concern for all hospitals, particularly in settings where resources are more limited.

The investigators aim to assess whether VL compared to DL results in more infants being intubated at the first attempt without physiological instability.

STUDY DESIGN A recent single centre study reported that that more newborn infants were successfully intubated at the first attempt when VL was used to indirectly view the airway compared to DL. This study was not large enough to determine the effect of VL on adverse effects that are seen commonly (e.g. desaturation) or more rarely (e.g. bradycardia, receipt of chest compressions or adrenaline, oral trauma) during intubation attempts.

For the current study, the investigators chose a stepped-wedge cluster randomised controlled design, where the participating centre, rather than the individual infant, will be the unit of randomisation. This design has been found appropriate to test the effects of an intervention that encompasses a behavioural aspect and to implement interventions while studying them at the same time. In this study, all centres will begin in the "control group"; where clinicians will routinely attempt intubation with DL, as is their usual practice. At specified intervals, centres will be randomly assigned to cross over to the "intervention group", where clinicians will routinely attempt intubation with VL. All participating centers will have included patients in both arms by the end of the study.

SAMPLE SIZE ESTIMATION To determine the intra-cluster correlation (that means the correlation between two observations from the same centre), the investigators used the dataset of the MONITOR trial that included infants from 7 delivery rooms worldwide. In this trial, the intra-cluster correlation for intubation in the delivery room was reported as 0.1.

This complete stepped-wedge cluster-randomized design includes 21 time periods (including the baseline) and 20 centres that will be including patients, with each randomised to a unique sequence. Each time period lasts a fortnight. Each time period, 1 centre will switch their treatment from DL to VL. With all centres including 2 patients each time period, 42 patients will be included per centre which will provide a total sample size of 840 patients.

Assuming a control proportion of 0.4, this sample will achieve 90% power (0.9091) to detect a treatment proportion of 0.55, assuming a conservative ICC of 0.05. The power is not very sensitive to ICC values up to 0.1 (power of >90% to detect difference 40% versus 56%). The test statistic used is the two-sided Wald Z-Test.

TREATMENT OF SUBJECTS

DIRECT LARYNGOSCOPY (DL, control period) At the start of the study, clinicians at participating centres will attempt intubation using a standard laryngoscope to perform DL as is their normal practice.

VIDEO LARYNGOSCOPY (VL, intervention period) For each centre, a lot will be drawn which indicates the month in which endotracheal intubation will be routinely attempted with VL rather than DL. In the month before the switch, centres will be provided with a C-MAC VL by the manufacturers, Karl Storz-Endoskop (Tuttlingen, Germany). The system will be provided on loan for the duration of the study and will consist of an 8" high-definition monitor with connecting cable and reusable straight Miller type blades size 0 and size 1. The equipment will be demonstrated by representatives from Karl Storz, and clinicians who intubate babies at participating hospitals will be encouraged to practice with the equipment on mannequins. We will have an virtual meeting with each centre in the week before they are due to switch to review the protocol, data collection and to answer any queries that they may have.

All other procedures in the delivery room and NICU will be performed according to international and local guidelines. All other aspects of the approach to intubation at the participating centre are at the discretion of the local clinicians and should remain the same for the duration of the study; e.g.:

* The drugs used before intubation attempts (e.g. opiate, atropine, curare-like drug)
* The route by which intubation is usually attempted (i.e. oral or nasal)
* Whether they use a stylet is routinely used
* Whether supplemental oxygen is given during attempts

ELIGIBILITY:
Inclusion Criteria:

* Infants of any gestational age in whom endotracheal intubation is attempted can be included in this study once there is parental consent to the use their infant's data.

Exclusion Criteria:

* Infants will be excluded if parents do not consent for their infants' data to be used.

Ages: 0 Minutes to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 840 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2025-12-13 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Successful intubation at the first attempt without physiologic instability | At 5 minutes from the start of the intubation attempt
  Successful intubation at the first attempt without physiologic instability where:
  1. an intubation attempt is defined as the introduction of the laryngoscope blade into the mouth, whether or not an attempt is made to pass an endotracheal tube (ETT);
  2. success is determined by detection of exhaled carbon dioxide (CO2) or with clinical signs (auscultation of breath sounds, condensation in the ETT);
  3. physiologic instability is defined as a fall in oxygen saturation (SpO2) of > 20% from the pre-attempt value or heart rate (HR) < 100 beats per minute (bpm) during the attempt

SECONDARY OUTCOMES:
Successful intubation at the first attempt | At 5 minutes from the start of the intubation attempt
  Successful intubation at the first attempt where:
  1. an intubation attempt is defined as introduction of the laryngoscope blade into the mouth, whether or not an attempt is made to pass an ETT;
  2. success is determined with exhaled CO2 or clinical signs (auscultation of breath sounds, condensation in the ETT)
Physiologic instability during the first intubation attempt | At 5 minutes from the start of the intubation attempt
  Fall in SpO2 > 20% from the pre-attempt value or HR < 100bpm during the first intubation attempt
Lowest SpO2 (%) measured with pulse oximetry during the procedure | At 5 minutes from the start of the intubation attempt
  Lowest oxygen saturation SpO2 (%) measured with pulse oximetry during the procedure
Lowest heart rate (HR) during the procedure | At 5 minutes from the start of the intubation attempt
  Lowest heart rate (HR) during the procedure
Number of intubation attempts taken to intubate successfully | At 30 minutes from the start of the intubation attempt
  Number of intubation attempts taken to intubate successfully
Total laryngoscopy time to successful intubation | At 30 minutes from the start of the intubation attempt
  Total laryngoscopy time to successful intubation defined as the sum of the duration of all intubation attempts (defined as the interval from the introduction of the laryngoscope blade into the mouth to its removal), measured in seconds
Number of participants successful intubated with assigned device | At 30 minutes from the start of the intubation attempt
  Number of participants successful intubated with assigned device
Number of participants reported by clinicians to have oral trauma within 1 hour of the intubation attempt | At 1 hour from the start of the intubation attempt
  Number of participants reported by clinicians to have oral trauma within 1 hour of the intubation attempt
Number of participants given adrenaline (IV or via ETT) within an hour of the intubation attempt | At 1 hour from the start of the intubation attempt
  Number of participants given adrenaline (IV or via ETT) within an hour of the intubation attempt
Number of participants given chest compressions within one hour of the intubation attempt | At 1 hour from the start of the intubation attempt
  Number of participants given chest compressions within one hour of the intubation attempt

CONTACTS AND LOCATIONS:
Locations (18):
- Croatia (2):
  - Clinical Hospital Centre, Rijeka
  - Clinical Hospital "Holy Spirit", Zagreb
- Czechia (3):
  - University Hospital Brno, Brno
  - General University Hospital, Prague
  - Institute for Mother and Child Care, Prague
- Aristotle University of Thessaloniki, Thessaloniki, Greece
- Second Semmelweiss University, Budapest, Hungary
- University of Padova, Padua, Italy
- Oslo University Hospital, Oslo, Norway
- Poland (5):
  - Medical University of Gdańsk, Gdansk
  - Medical University of Silesia, Katowice
  - Poznań University of Medical Sciences, Poznan
  - Provincial Hospital No. 2, Rzeszów
  - Wrocław Medical University, Wroclaw
- Romania (2):
  - Clinical County Emergency Hospital, Sibiu
  - George Emil Palade University, Tărgu Mures
- University and Polytechnic Hospital La Fe, Valencia, Spain
- Bukovinian State Medical University, Chernivtsi, Ukraine

IPD SHARING:
Plan to Share IPD: Yes
Reasonable requests for IPD will be considered by the investigators
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 2 years
Access Criteria: Reasonable requests for IPD will be considered by the investigators

REFERENCES:
- [Background] Geraghty LE, Dunne EA, Ni Chathasaigh CM, Vellinga A, Adams NC, O'Currain EM, McCarthy LK, O'Donnell CPF. Video versus Direct Laryngoscopy for Urgent Intubation of Newborn Infants. N Engl J Med. 2024 May 30;390(20):1885-1894. doi: 10.1056/NEJMoa2402785. Epub 2024 May 5. PMID 38709215
- [Background] Sawyer T, Foglia EE, Ades A, Moussa A, Napolitano N, Glass K, Johnston L, Jung P, Singh N, Quek BH, Barry J, Zenge J, DeMeo SD, Brei B, Krick J, Kim JH, Nadkarni V, Nishisaki A; National Emergency Airway Registry for Neonates (NEAR4NEOS) investigators. Incidence, impact and indicators of difficult intubations in the neonatal intensive care unit: a report from the National Emergency Airway Registry for Neonates. Arch Dis Child Fetal Neonatal Ed. 2019 Sep;104(5):F461-F466. doi: 10.1136/archdischild-2018-316336. Epub 2019 Feb 22. PMID 30796059
- [Background] Singh N, Sawyer T, Johnston LC, Herrick HM, Moussa A, Zenge J, Jung P, DeMeo S, Glass K, Howlett A, Shults J, Barry J, Brei BK, Kim JH, Quek BH, Tingay D, Mehrem AA, Napolitano N, Nishisaki A, Foglia EE; National Emergency Airway Registry for Neonates (NEAR4NEOS). Impact of multiple intubation attempts on adverse tracheal intubation associated events in neonates: a report from the NEAR4NEOS. J Perinatol. 2022 Sep;42(9):1221-1227. doi: 10.1038/s41372-022-01484-5. Epub 2022 Aug 18. PMID 35982243
- [Background] Foglia EE, Ades A, Sawyer T, Glass KM, Singh N, Jung P, Quek BH, Johnston LC, Barry J, Zenge J, Moussa A, Kim JH, DeMeo SD, Napolitano N, Nadkarni V, Nishisaki A; NEAR4NEOS Investigators. Neonatal Intubation Practice and Outcomes: An International Registry Study. Pediatrics. 2019 Jan;143(1):e20180902. doi: 10.1542/peds.2018-0902. Epub 2018 Dec 11. PMID 30538147
- [Background] American Academy of Pediatrics/American Heart Association. Textbook of Neonatal Resuscitation (8th ed, June 2021), editors Weiner GM, Zaichkin J. AAP, Elk Grove, IL USA.